CLINICAL TRIAL: NCT01148875
Title: Finding the M.I.N.C. for Mammography Maintenance
Brief Title: Mammography Reminders for Encouraging Women to Undergo Regular Mammography Screenings for Breast Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UNC-03-2104; R01CA105786 (NIH); P30CA016086 (NIH); CDR0000438777 (Other: PDQ number)
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; mammography adherence; non-adherent
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Mammography appointment reminders; telephone counseling — Women randomly assigned to UCR, EAPR, ELR; repeated 4 times at yearly intervals. Using claims data, supplemented by self-report, verified if women had recent mammograms. Women who remained non-adherent after reminders received Barriers-Specific Telephone Counseling Call, or an enhanced call including focus on either positive or negative consequences of getting/not getting mammograms. Prior to calls, women in each of the three phone counseling groups received priming letters to prime them to process information in the call. Priming letters should prepare women to process information from subsequent counseling calls more deeply by focusing on the positive or negative consequences of getting/not getting mammograms or on identifying and overcoming their own barriers to being screened.
  Other Names: Usual Care Reminder(UCR); Enhanced Automated Phone Reminder (EAPR); Enhanced Letter Reminder (ELR); Priming Letter (PL); BarriCall; BarriConCall+; BarriConCall-

SUMMARY:
RATIONALE: Mammography reminders may encourage women to undergo regular mammography screenings for breast cancer.

PURPOSE: This randomized clinical trial is studying three different mammography reminder interventions to compare how well they work in encouraging women to undergo regular mammography screenings for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of mammography reminder interventions using usual care reminder vs enhanced automated phone reminder vs enhanced letter reminder in increasing the proportion of women who undergo annual mammograms as recommended by medical organizations.
* Compare the impact of alternative delivery channels (mail vs automated phone reminders) and enhanced messages in facilitating maintenance of mammography in these participants.
* Determine the incremental benefit of adding a consequence elaboration component to barriers-specific telephone counseling in encouraging these participants to regain adherence to mammography.
* Determine the minimum intervention needed for change to ensure annual mammography and maintenance in participants.

OUTLINE: This is a randomized, controlled study. Participants are randomized to 1 of 3 arms.

* Arm I: Participants receive a usual care mammography reminder by telephone annually for 4 years.
* Arm II: Participants receive an enhanced automated phone mammography reminder annually for 4 years.
* Arm III: Participants receive an enhanced letter mammography reminder annually for 4 years.

Insurance claims reports and patients' self reports as to whether or not they subsequently underwent mammography are examined. Patients who do not undergo mammography within 6 months after receiving a reminder are further randomized to 1 of 4 arms.

* Arm I: Participants receive no further reminders until the next annual reminder.
* Arm II: Participants receive an enhanced Barriers-Specific Counseling Call (BarriConCall) annually for 4 years that focuses on positive consequences of undergoing mammography.
* Arm III: Participants receive an enhanced BarriConCall annually for 4 years that focuses on negative consequences of not undergoing mammography.
* Arm IV: Participants receive a standard barrier call (BarriCall) annually for 4 years.

PROJECTED ACCRUAL: A total of 4,040 participants (1,000 for usual care mammography reminder; 1,520 for enhanced automated phone mammography reminder; and 1,520 for enhanced letter mammography reminder) will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

1. Women members of The North Carolina Teachers' and State Employees' Comprehensive Major Medical Plan (SHP)
2. Age 40-75
3. Enrolled with the SHP for at least 24 months, not covered by COBRA or Medicare primary
4. Based on claims data, women will have had their last mammogram 6-8 months ago so reminders will arrive 2 months prior to due date for next mammogram.

Exclusion criteria:

1. Unable to speak and understand English. We lack the resources to adapt the intervention appropriate for non-English speakers. Moreover, we do not know if the interventions lend themselves to cultural translation. We regard this as a next logical research activity.
2. Have breast cancer or have some other illness that precludes participation. Women diagnosed with breast cancer before the study are ineligible; their screening schedules are consistent with recommendations for the general population. However, if women develop breast cancer during the study, we would ask them a reduced set of questions.

We selected age 75 as the upper limit, because there are too few women over age 75 to permit meaningful statistical analysis (<100 women in all). The SHP is largely a working population. We wish that it were possible both to include and analyze women older than age 75. This is a limitation of the population we have selected.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women members of The North Carolina Teachers' and State Employees' Comprehensive Major Medical Plan (SHP) who are age 40-75. They must be enrolled with the SHP for at least 24 months, not covered by COBRA or Medicare primary. Based on claims data, women will have had their last mammogram 6-8 months ago.
Sampling Method: Probability Sample
Enrollment: 3547 (Actual)
Dates: Start 2004-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Mammography Adherence | 12 months
  The primary study objective was to identify the minimal intervention needed for sustained mammography adherence over 4 years. Average cumulative number of days non-adherent to mammography over 4 years based on annual screening guidelines. Claims data (monthly mammography claims information were reviewed to determine women's adherence status) and self-report (during annual telephone interviews, women were asked to confirm dates of their most recent and prior mammograms, based on claims data) were used to determine dates of screening.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K. Rimer, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center

REFERENCES:
- [Background] Lipkus, I.M., Klein, W.M.P., Skinner, C.S., Rimer, B.K. (2005) Breast Cancer Risk Perceptions and Breast Cancer Worry: What Predicts What? Journal of Risk Research, 8(5): 439-452.
- [Background] Rimer BK, Gierisch JM. Public education and cancer control. Semin Oncol Nurs. 2005 Nov;21(4):286-95. doi: 10.1016/j.soncn.2005.06.003. PMID 16293517
- [Background] Rimer, B.K. and Kreuter, M.W. (2006). Advancing Tailored Health Communication: A Persuasion and Message Effects Perspective. Journal of Communication, (56): S184-S201.
- [Background] Gierisch JM, Reiter PL, Rimer BK, Brewer NT. Standard definitions of adherence for infrequent yet repeated health behaviors. Am J Health Behav. 2010 Nov-Dec;34(6):669-79. doi: 10.5993/ajhb.34.6.4. PMID 20604693
- [Result] DeFrank JT, Bowling JM, Rimer BK, Gierisch JM, Skinner CS. Triangulating differential nonresponse by race in a telephone survey. Prev Chronic Dis. 2007 Jul;4(3):A60. Epub 2007 Jun 15. PMID 17572964
- [Result] O'Neill SC, Bowling JM, Brewer NT, Lipkus IM, Skinner CS, Strigo TS, Rimer BK. Intentions to maintain adherence to mammography. J Womens Health (Larchmt). 2008 Sep;17(7):1133-41. doi: 10.1089/jwh.2007.0600. PMID 18657041
- [Result] DeFrank JT, Rimer BK, Gierisch JM, Bowling JM, Farrell D, Skinner CS. Impact of mailed and automated telephone reminders on receipt of repeat mammograms: a randomized controlled trial. Am J Prev Med. 2009 Jun;36(6):459-67. doi: 10.1016/j.amepre.2009.01.032. Epub 2009 Apr 11. PMID 19362800
- [Result] Gierisch JM, O'Neill SC, Rimer BK, DeFrank JT, Bowling JM, Skinner CS. Factors associated with annual-interval mammography for women in their 40s. Cancer Epidemiol. 2009 Jul;33(1):72-8. doi: 10.1016/j.cdp.2009.03.001. Epub 2009 May 29. PMID 19481879
- [Result] Gierisch JM, DeFrank JT, Bowling JM, Rimer BK, Matuszewski JM, Farrell D, Skinner CS. Finding the minimal intervention needed for sustained mammography adherence. Am J Prev Med. 2010 Oct;39(4):334-44. doi: 10.1016/j.amepre.2010.05.020. PMID 20837284
- [Result] Gierisch JM, Earp JA, Brewer NT, Rimer BK. Longitudinal predictors of nonadherence to maintenance of mammography. Cancer Epidemiol Biomarkers Prev. 2010 Apr;19(4):1103-11. doi: 10.1158/1055-9965.EPI-09-1120. Epub 2010 Mar 30. PMID 20354125
- [Result] Mier N, Ory MG, Toobert DJ, Smith ML, Osuna D, McKay JR, Villarreal EK, DiClemente RJ, Rimer BK. A qualitative case study examining intervention tailoring for minorities. Am J Health Behav. 2010 Nov-Dec;34(6):822-32. PMID 20604705
- [Result] O'Neill SC, Lipkus IM, Gierisch JM, Rimer BK, Bowling JM. It's the amount of thought that counts: when ambivalence contributes to mammography screening delay. Womens Health Issues. 2012 Mar;22(2):e189-94. doi: 10.1016/j.whi.2011.08.008. Epub 2011 Nov 3. PMID 22055988